CLINICAL TRIAL: NCT01959971
Title: A Phase 1 Study of the Effects of Subcutaneous Doses of Alirocumab on Lipid and Lipoprotein Metabolism in Adults With Mildly Elevated LDL-Cholesterol
Brief Title: Effect of Alirocumab on Lipid Metabolism in Adults With Elevated LDL-Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PDY13670; U1111-1141-4567 (Other: UTN)
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Intervention Model Description: Single-sequence crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo - Alirocumab (Experimental): Injection through subcutaneous (SC) administration, placebo for 4 weeks then, alirocumab for 10 weeks
  Interventions: Drug: alirocumab; Drug: Placebo

INTERVENTIONS:
Drug: alirocumab — Pharmaceutical form:Solution for injection
  Route of administration: Subcutaneous
  Other Names: SAR236553; REGN727; Praluent
Drug: Placebo — Pharmaceutical form:Solution for injection
  Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To assess the effects of subcutaneous (SC) doses of alirocumab on the elimination (measured by Fractional Clearance Rate (FCR)) of apolipoprotein B (apoB) in low density lipoprotein (LDL) in adults with mildly elevated LDL-cholesterol (LDL-C).

Secondary Objectives:

To assess the effects of SC doses of alirocumab on:

* Various parameters of the metabolism and turnover in plasma of different lipoproteins
* Plasma lipids concentration: total cholesterol, high density lipoprotein cholesterol (HDL-C), triglycerides, low density lipoprotein cholesterol (LDL-C), apoB, lipoprotein(a) (Lp(a))
* Lipoprotein particle size profile
* PCSK9 (free and total) concentrations in serum To assess safety and tolerability of alirocumab. To assess emergence of anti-alirocumab antibodies. To document serum alirocumab concentrations.

DETAILED DESCRIPTION:
Total duration of the study per subject is 26 weeks, including a screening period of ≤ 4 weeks, placebo treatment period of 4 weeks, alirocumab treatment period of 10 weeks, and a follow up period of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

Generally healthy; LDL-C level in serum or plasma ≥ 100 mg/dL and < 190 mg/dL at Screening.

Exclusion criteria:

* LDL-C ≥ 160 mg/dL at Screening if more than 2 major Coronary Heart Disease risk factors, as defined in National Cholesterol Education Program guidelines.
* Receiving treatment of any kind for hyperlipidemia within 6 weeks of enrollment.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percent change in Fractional Clearance Rate of apolipoprotein B (apoB) in Low Density Lipoproteins (pools/day) in plasma during alirocumab treatment | baseline and at 12 days after last dose of alirocumab

SECONDARY OUTCOMES:
Change in lipids turnover parameters measured in isolated Very Low Density Lipoproteins (VLDL), Intermediate Density Lipoproteins (IDL), Low Density Lipoproteins (LDL) and High Density Lipoproteins (HDL) | baseline and at 12 days after last dose of alirocumab
Change in post-heparin hepatic lipase and lipoprotein lipase activities | baseline and at 2 days after last dose of alirocumab
Change in lipids and apolipoproteins in plasma lipids panel | baseline and at 2 days and at 11 days after last dose of alirocumab
Assessment of Lipoprotein particle size profiles | baseline and at 2 days and at 11 days after last dose of alirocumab
Assessment of serum concentrations of PCSK9 | baseline and up to 2 weeks after last dose of alirocumab
Assessment of safety parameters (clinical laboratory, ECG, vital signs) | up to 10 weeks after last dose of alirocumab
Assessment of the serum concentration of alirocumab | baseline and up to 2 weeks after last dose of alirocumab
Assessment of the serum concentration of anti-alirocumab antibodies | baseline and up to 10 weeks after last dose of alirocumab

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, New York, New York, United States

REFERENCES:
- [Result] Reyes-Soffer G, Pavlyha M, Ngai C, Thomas T, Holleran S, Ramakrishnan R, Karmally W, Nandakumar R, Fontanez N, Obunike J, Marcovina SM, Lichtenstein AH, Matthan NR, Matta J, Maroccia M, Becue F, Poitiers F, Swanson B, Cowan L, Sasiela WJ, Surks HK, Ginsberg HN. Effects of PCSK9 Inhibition With Alirocumab on Lipoprotein Metabolism in Healthy Humans. Circulation. 2017 Jan 24;135(4):352-362. doi: 10.1161/CIRCULATIONAHA.116.025253. Epub 2016 Dec 16. PMID 27986651